CLINICAL TRIAL: NCT00430976
Title: Exercise, Executive Processes and the Aging Brain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IA0101; 5R01AG021188-03 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2008-08

CONDITIONS: Cognition; Aging
Keywords: psychomotor function; neuromuscular system; memory; brain electrical activity; Mental Processes
MeSH Terms: interventions — Motion

INTERVENTIONS:
Behavioral: Minds in Motion

SUMMARY:
The purpose of this study is to assess the effect of aerobic exercise on the brain and cognition through the measurement of neuroelectric and behavioral indices of executive control cognitive function in older adults.

DETAILED DESCRIPTION:
The aim of this research is to gain a better understanding of factors that relate to the increased health and effective functioning of older adults. Specifically, efficiency of psychomotor performance declines with advancing age leading to profound effects on older adults' quality of life. For this reason, researchers have focused on the influence that individual lifestyle habits have on the aging process. One lifestyle choice that has been found to positively contribute to the efficiency of older adults' psychomotor performance is cardiovascular exercise. This relationship appears to be especially significant when older adults are challenged with more complex or effortful tasks. Previous research has led investigators to believe that aging has a specific, rather than generalized, impact on cognitive functioning. Also, prolonged participation in cardiovascular exercise has been found to maintain the cognitive functioning critical for healthy aging.

Therefore, the purpose of this research is to examine the role of an organized 6-month cardiovascular exercise intervention trial on electrocortical (event-related brain potential) and behavioral measures (reaction time) of executive control. In addition, a non-cardiovascular exercise control group that participates in a 6-month stretching and toning program will be used for comparison. Participants will be measured before and after exercise training during engagement in several tasks designed to elicit different executive functions (e.g., discrimination, task switching, inhibition). Each task also contains a non-executive condition that will be used for comparison to examine the specificity of exercise participation of cognitive functioning. A secondary aim of this project is to determine the effects of an acute bout of exercise on cognitive functioning. Both groups will participate in several bouts of exercise followed by immediate measurement on the tasks outlined above to determine whether acute exercise has beneficial effects on executive processes. The significance of this research may include the increased understanding of factors related to the amelioration of age-related decrements in central nervous system functioning and recommendations for the maintenance of cognitive health during the later stages of life.

ELIGIBILITY:
Inclusion Criteria:

* 60-74 years of age
* Sedentary (no physical activity in 6 last months)
* Capable of performing exercise
* Personal physician's examination and consent to participate in testing and exercise or control intervention
* Successful completion of graded exercise test without evidence of cardiac abnormalities or responses
* Adequate performance on the Mental Status measure
* Corrected (near and far) acuity 20/40 or better
* Initial depression score on GDS below clinical level
* Not previously committed to leaving the Champaign County area for more than 1 month during the intervention period

Exclusion Criteria:

* Below 60 years of age
* Regular self-reported physical activity (2 times per week) in last six months
* Any physical disability that prohibits mobility (walking), stretching etc.
* Non-consent of physician
* Evidence of abnormal cardiac responses or conditions during graded exercise testing
* Three or more errors on the Mental Status measure
* Corrected (near and far) acuity of greater than 20/40
* Depression score on GDS indicative of clinical depression
* Committed to leaving the Champaign County area for longer than 1 month during the intervention period

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Changes in event-related brain potentials
reaction time
response accuracy

SECONDARY OUTCOMES:
aerobic fitness

CONTACTS AND LOCATIONS:
Overall Officials: Charles H. Hillman, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Background] Themanson JR, Hillman CH, Curtin JJ. Age and physical activity influences on action monitoring during task switching. Neurobiol Aging. 2006 Sep;27(9):1335-45. doi: 10.1016/j.neurobiolaging.2005.07.002. Epub 2005 Aug 15. PMID 16102874
- [Background] Hillman CH, Motl RW, Pontifex MB, Posthuma D, Stubbe JH, Boomsma DI, de Geus EJC. Physical activity and cognitive function in a cross-section of younger and older community-dwelling individuals. Health Psychol. 2006 Nov;25(6):678-687. doi: 10.1037/0278-6133.25.6.678. PMID 17100496
- [Background] Hillman CH, Kramer AF, Belopolsky AV, Smith DP. A cross-sectional examination of age and physical activity on performance and event-related brain potentials in a task switching paradigm. Int J Psychophysiol. 2006 Jan;59(1):30-9. doi: 10.1016/j.ijpsycho.2005.04.009. PMID 16413382